CLINICAL TRIAL: NCT00566462
Title: Assessment of Perampanel (E2007) on Synaptic Dopamine in Mild-moderate PD Patients: A Pilot Study With [^123I]-IBZM SPECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-226
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- perampanel (Experimental)
  Interventions: Drug: perampanel
- 1 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: perampanel — 2 mg/d for 14 days followed by 4 mg/d for 14 days
  Arms: perampanel
Drug: placebo — Matching placebo for for 14 days followed by 4 mg/d for 14 days
  Arms: 1

SUMMARY:
This is a two-arm, double-blind, placebo-controlled study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients with idiopathic PD fulfilling the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) diagnostic criteria, with a good response to levodopa. The requirement in the UKPDSBB Step 2 for prior brain imaging is at the discretion of the investigator.

   * Clinical diagnosis of idiopathic Parkinson's disease (patients must have at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia)
   * Hoehn and Yahr Stage II to IV.
   * Treatment with monotherapy of levodopa plus an aromatic acid decarboxylase inhibitor (carbidopa). The carbidopa/levodopa medication should be taken at least two times daily (excluding the bedtime/night time dose) up to a maximum of eight doses daily (including the bedtime/night time dose).
   * Intermittent use of either liquid forms of levodopa or subcutaneous apomorphine is permitted.
   * Age >30 years of age
   * Women who are incapable of bearing children (e.g., clinically assessed as infertile, including surgically sterile) or who are practicing effective contraception (e.g., abstinence, intrauterine device or barrier method plus hormonal method).

   Postmenopausal women may be recruited but must be amenorrheic for at least 1 year to be considered. Women must have a negative serum beta-human chorionic gondotrophin (β-HCG) test at the Screening Visit and a negative urine pregnancy test prior to radiotracer administration on the day of each SPECT scanning session. Women must also be willing to remain on their current form of contraception for the duration of the study.
2. In the investigator's opinion, patients are able to complete the study and are capable of giving full written informed consent.

EXCLUSION CRITERIA:

Patients with any one of the following will be excluded:

1. Inability or unwillingness to undergo SPECT or other study procedures
2. Pregnant or lactating women
3. Atypical or drug-induced PD
4. Current treatment with dopamine agonists, MAO or COMT inhibitors, anticholinergics
5. Patients with a past (within 1 year) or present history of psychotic symptoms requiring antipsychotic treatment. Patients may be taking antidepressant medication, however, the dose must be stable for 4 weeks prior to the Baseline Visit. Use of antipsychotic medication including clozapine and quetiapine is prohibited, even if the indication is for movement disorders.
6. Current or prior treatment (within 4 weeks prior to Baseline Visit) with pergolide, tolcapone, methyldopa, budipine, reserpine, seroquel, or the herbal dopamine agonist, Mucuna Pruriens
7. Patients with current or prior treatment (within 4 weeks prior to the Baseline Visit) with medication known to induce the enzyme cytochrome P450 3A4
8. Use of an investigational product within 4 weeks prior to randomization or patients who have participated in a previous study with perampanel
9. Patients with a past or present history of drug or alcohol abuse as per Diagnostic and Statistical Manual - 4th edition (DSM IV) criteria
10. Dementia (as defined by a MMSE score of ≤ 24) and/or fulfilling the criteria for dementia due to PD (as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association - 4th Edition)
11. Clinically significant unstable medical or psychiatric illness
12. Presence of physical, mental, or social condition that precludes informed consent or interferes with careful follow-up
13. Past (within 1 year) or present history of suicidal ideation or suicide attempts
14. Elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of normal (ULN)
15. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastrointestinal, haematological, endocrine, or metabolic systems that might complicate assessment of the tolerability of the study medication
16. Evidence of significant active hematological disease: white blood cell (WBC) count ≤ 2500/μL; absolute neutrophil count ≤ 1000/μL
17. Patients with previous stereotactic surgery (eg, pallidotomy) for Parkinson's disease or with planned stereotactic surgery during the study period
18. Patients receiving or planning to receive (within 3 months) deep brain stimulation
19. Patients with conditions affecting the peripheral or central sensory system unless related to Parkinson's disease (such as mild sensory or pain syndromes limited to "OFF" periods) that could interfere with the evaluation of any such symptoms caused by the study drug
20. Patients with any condition that would make the patient, in the opinion of the investigator, unsuitable for the study
21. Patients with clinically significant ECG abnormality, including prolonged QTc (defined as QTc > 450 msec)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Cole, PhD, MD, Study Director — Eisai Inc.
Locations (3):
- United States (3):
  - Kenneth Marek, New Haven, Connecticut
  - Molecular NeuroImaging, LLC, New Haven, Connecticut
  - inVentiv, The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel: A single dose carbidopa/levodopa (37.5mg/150mg PO) challenge at Baseline, followed by one 2-mg tablet/day PO of Perampanel for 14 days, then two 2-mg tablets/day (4-mg/day)PO of Perampanel for 14 days, followed by a single dose carbidopa/levodopa (37.5mg/150mg PO) challenge after 4 weeks.
- Placebo: A single dose carbidopa/levodopa (37.5mg/150mg PO) challenge at Baseline, followed by one 2-mg tablet/day PO of perampanel-matched placebo for 14 days, then two 2-mg tablets/day (4-mg/day)PO of perampanel-matched placebo for 14 days, followed by a single dose carbidopa/levodopa (37.5mg/150mg PO) challenge after 4 weeks.
Period: Overall Study
Arm/Group | Perampanel | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Striatal [^123I]-Iodobenzamine (IBZM_ Binding Following a Single Dose Carbidopa/Levodopa Challenge for 15-hours at Baseline and Week 4
Time Frame: Baseline and Week 4
Population: No data was collected because the study was terminated at the sponsor request due to low enrollment.
Arm/Group | Perampanel | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Caudate and Putamen [^123I]-IBZM Binding Following a Single Dose Carbidopa/Levodopa Challenge for 15-hours at Baseline and Week 4
Time Frame: Baseline and Week 4
Population: No data was collected because the study was terminated at the sponsor request due to low enrollment.
Arm/Group | Perampanel | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Perampanel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=1) | Placebo (N=0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Frontal Headache (Nervous system disorders) | 1 | 0
Sore Tongue (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated at the sponsor request after only 1 subject was enrolled and completed the study and therefore the data is limited. Similiar research in this area have required a minimum of 5-6 completers to develop a valid analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other